CLINICAL TRIAL: NCT03553550
Title: Role of Circulating Tumor DNA (ctDNA) From LIquid Biopsy in Early Stage NSCLC Resected Lung Tumor Investigation
Acronym: LIBERTI
Status: Terminated | Type: Observational
Why Stopped: Enrollment futility
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-010
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue - The participant will be asked to provide a tissue sample collected during a clinically-indicated surgery for NSCLC. This sample will be divided and put on to slides to be seen under a microscope. The slides will be stored at the ALCMI Biorepository for future lung cancer research purposes. The slides may be selected to study circulating tumor cells (cells from the tumors that circulate in the bloodstream) and their patterns.
  Peripheral blood - The blood will be sent to a company named, IniVata, to study the changes in circulating tumor cells (cells from the tumors that circulate in the bloodstream) as well as DNA (parts of the cell that carry genetic information) most often seen in NSCLC. We expect the research testing to consume the entire blood specimen. However, if any residual blood specimen remains, it will be stored at IniVata however, it cannot be used without ALCMI's permission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biospecimen collection — Peripheral blood collection Archival tissue collection

SUMMARY:
The purpose of this research study is to learn more about changes in cell-free tumor DNA in blood samples, also known as a liquid biopsy, as they relate to treatment and response to treatment.

DETAILED DESCRIPTION:
Every type of cancer is associated with changes in genes and protein structure or function in the body known as "biomarkers". These biomarkers can help diagnose cancer, as well as to track the disease and response to treatment. Over the last 10 years, technology has led to the identification of many cancer biomarkers; the use of cancer biomarkers has become an important part in the treatment and management of cancer.

For solid tumors, biomarker testing is usually done on the tumor tissue from a biopsy or surgery. Although testing tumor tissue provides a lot of information, there are some challenges with the process. First, tumor cells can be different even within small tumors. To overcome this, the pathologist (doctor that examines tumor tissue) needs to test cells from different parts of the tumor. Often, there may not be enough of the tissue to test for biomarkers. In addition, tumor cells change when the patient undergoes treatment and there might be a need to repeat biopsies. Sometimes it may not be possible to repeat a biopsy to study the changes in biomarkers because some patients cannot have a repeat biopsy done safely.

There are many advantages to tracking biomarkers in the blood instead of on tissue. We can study changes in biomarkers more often (because it is a blood draw), and therefore will be able to determine how your treatment is working, learn if the cancer is coming back, or find drugs that may target the changed tumor cells.

The purpose of this research study is to learn more about changes in cell-free tumor DNA in blood samples, also known as a liquid biopsy, as they relate to treatment and response to treatment. Cell-free tumor DNA is genetic material that is released into your bloodstream from tumor cells as they die. Genes are a unique combination of molecules (called DNA) that are found in all human cells. In some cases, these genes may be changed in cancer and tumor cells. These changes, or tumor markers are substances produced by cancer cells that are found in the blood, body fluids or tissues, and may be made of DNA, RNA, proteins, cells or components of cells. In the future, the "markers" may help doctors decide which treatments could be most beneficial for NSCLC. Tumor markers may be used to help predict a response to certain cancer treatments and to check how the patiet's type of cancer responds to the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years and over
2. Planned surgical resection of NSCLC, stage IB ≥ 4 cm, II or IIIA according to the 8th edition of TNM classification16.

   1. Cohort #1: Neoadjuvant Therapy - For patients who will receive neoadjuvant therapy, enrollment occurs prior to the initiation of treatment. Patients undergoing neoadjuvant therapy who achieved tumor reduction, are eligible based on baseline radiographic staging.
   2. Cohort #2: Pre-Surgery - For patients identified prior to planned surgical resection, enrollment occurs within 30 days of the planned surgery. Eligibility is based on surgical pathology.
   3. Cohort #3: Post-Surgery - For patients identified post-surgical resection, enrollment occurs prior to the initiation of adjuvant therapy. Eligibility is based on surgical pathology.
3. Patients with positive margins and those requiring adjuvant radiation therapy are eligible.
4. Patients with a secondary malignancy that was treated with curative intent and without evidence of relapse for at least 5 years.
5. Willingness to undergo all study collection procedures and follow up.
6. Provision of written informed consent

Exclusion Criteria:

1. Male or female aged less than 18 years
2. NSCLC disease other than stated above
3. Patients with a secondary malignancy that was not treated with curative intent or has had a disease relapse in the past 5 years.
4. Unwilling to undergo all study collection procedures and follow up.
5. Unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Stage IB, II or IIIA NSCLC that have a planned surgery to treat their cancer.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
To correlate the presence of ctDNA following complete surgical resection with disease-free survival. | June, 2023
  Correlation between ctDNA after surgery and disease-free survival, defined as the time from surgical resection to the earliest event defined as disease recurrence, death or new lung cancer.

SECONDARY OUTCOMES:
To evaluate the relation between changes in ctDNA during surveillance and tumor relapse | June, 2023
  Evaluate the changes in ctDNA after complete resection at pre-specified intervals and correlate the presence of ctDNA with overall survival.

OTHER OUTCOMES:
Overall survival | June, 2023
  Evaluate the effect of adjuvant therapy on the ctDNA levels and tumor relapse, ct DNA alterations during the follow-up and concordance between mutations detected in the operative specimens and ct DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, MD, Principal Investigator — Washington University School of Medicine
Locations (6):
- United States (6):
  - Northside Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - St. Louis Cancer Care, Bridgeton, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
no IPD plan created as no individual participate data will be available to other researchers.